CLINICAL TRIAL: NCT04893343
Title: Antibiotic Use in a Neonatal Intensive Care Unit Practicing Integrative Medicine
Status: Completed | Type: Observational
Sponsor: ARCIM Institute Academic Research in Complementary and Integrative Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: NEO_01
Record Dates: First submitted 2021-04-26; First posted 2021-05-19 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Neonatal Infection
Keywords: Neonatal infection; Neonatal sepsis; Antibiotic prescribing; Antibiotic stewardship
MeSH Terms: conditions — Neonatal Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neonatal infection with antibiotics: In-patient neonates with ICD-10 infectious disease diagnosis, treated with antibiotics
  Interventions: Other: Antibiotic treatment
- Neonatal infection without antibiotics: In-patient neonates with ICD-10 infectious disease diagnosis, treated without antibiotics
  Interventions: Other: No antibiotic treatment

INTERVENTIONS:
Other: Antibiotic treatment — Antibiotic treatment
  Groups: Neonatal infection with antibiotics
Other: No antibiotic treatment — No antibiotic treatment
  Groups: Neonatal infection without antibiotics

SUMMARY:
The goal of this study is to describe the antibiotic use in a neonatal intensive care unit (NICU) in Germany that is practising integrative medicine. The investigators will review hospital records to find out how often and how long antibiotics were given to newborns; compare antibiotic use to other NICU in the same area; describe how sick infected newborns were (comparing those treated with or without antibiotics); and describe which anthroposophic medicines were used, how often and if there were safety problems.

DETAILED DESCRIPTION:
A retrospective study, analysing antibiotic use in a level 2 neonatology intensive care unit (NICU) in Germany over a 4-year period from 2014 to 2017. The study will analyse frequency of antibiotic prescribing; compare antibiotic use to other level 2 NICU; compare clinical and laboratory parameters among neonates with infectious disease diagnosis managed with or without antibiotics; use and tolerability of anthroposophic medicinal products.

ELIGIBILITY:
Inclusion Criteria:

* Admission to neonatal intensive care unit

Exclusion Criteria:

* None

Ages: 0 Days to 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonates (aged 0 to 30 days) who are hospitalized for neonatal infection.
Sampling Method: Non-Probability Sample
Enrollment: 246 (Actual)
Dates: Start 2021-06-15 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Antibiotic prescription rate | January 1, 2014 to December 31, 2017
  Number of antibiotic treatment days per 100 hospital days

SECONDARY OUTCOMES:
Antibiotic use compared to other level 2 NICU in same geographic area | January 1, 2014 to December 31, 2017
  Proportion of neonates having received any antibiotic, compared to proportion in other level 2 NICU in the same geographic area
Antibiotic type | January 1, 2014 to December 31, 2017
  Types of antibiotics used, frequency of use per antibiotic type
Antibiotic treatment duration | January 1, 2014 to December 31, 2017
  Mean treatment duration and distribution among recommended therapy durations: 48 hours, 5 days and 7-10 days durations
Clinical and laboratory parameters in neonates with infectious disease diagnosis: Premature rupture of membranes | January 1, 2014 to December 31, 2017
  Descriptive analysis of clinical and laboratory parameters in neonates with ICD-10 infectious disease diagnosis, treated with and without antibiotics. Here: Premature rupture of membranes >24h before birth
Clinical and laboratory parameters in neonates with infectious disease diagnosis: Mother group B streptococcus positive | January 1, 2014 to December 31, 2017
  Descriptive analysis of clinical and laboratory parameters in neonates with ICD-10 infectious disease diagnosis, treated with and without antibiotics. Here: Mother tested positive for group B streptococcus
Clinical and laboratory parameters in neonates with infectious disease diagnosis: Low birthweight | January 1, 2014 to December 31, 2017
  Descriptive analysis of clinical and laboratory parameters in neonates with ICD-10 infectious disease diagnosis, treated with and without antibiotics. Here: Neonates with low birthweight (< 2500 g)
Clinical and laboratory parameters in neonates with infectious disease diagnosis: pH umbilical artery at birth | January 1, 2014 to December 31, 2017
  Descriptive analysis of clinical and laboratory parameters in neonates with ICD-10 infectious disease diagnosis, treated with and without antibiotics. Here: pH of umbilical artery blood at birth
Clinical and laboratory parameters in neonates with infectious disease diagnosis: Infant fever on admission | January 1, 2014 to December 31, 2017
  Descriptive analysis of clinical and laboratory parameters in neonates with ICD-10 infectious disease diagnosis, treated with and without antibiotics. Here: Infant fever on admission (≥ 38.0° C)
Clinical and laboratory parameters in neonates with infectious disease diagnosis: CRP maximum value | January 1, 2014 to December 31, 2017
  Descriptive analysis of clinical and laboratory parameters in neonates with ICD-10 infectious disease diagnosis, treated with and without antibiotics. Here: Maximum value of C-reactive protein (mg/l)
Clinical and laboratory parameters in neonates with infectious disease diagnosis: Leukocyte count maximum value | January 1, 2014 to December 31, 2017
  Descriptive analysis of clinical and laboratory parameters in neonates with ICD-10 infectious disease diagnosis, treated with and without antibiotics. Here: Maximum value of leukocyte count (cells per liter)
Use of anthroposophic medications: medication names | January 1, 2014 to December 31, 2017
  Anthroposophic medications: names of the medications used
Use of anthroposophic medications: frequency of use | January 1, 2014 to December 31, 2017
  Anthroposophic medications: frequency of use per medication
Safety of anthroposophic medications: side effects | January 1, 2014 to December 31, 2017
  Recording of anthroposophic medication side effects
Safety of anthroposophic medications: adverse drug reactions | January 1, 2014 to December 31, 2017
  Recording of anthroposophic medication adverse drug reactions (ADR, in grades I-IV, ADR as % of prescriptions)

CONTACTS AND LOCATIONS:
Overall Officials: Jan Vagedes, Dr, Principal Investigator — Arcim Institute
Locations (1):
- Die Filderklinik, Filderstadt, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication
Time Frame: The data will be made available upon publication for a duration of three months.
Access Criteria: The data will be made available to researchers who provide a methodologically sound proposal for use in achieving the goals of the approved proposal.

REFERENCES:
- [Derived] Vagedes J, Huber BM, Islam MOA, Vagedes K, Kohl M, Schoen-Angerer TV. Antibiotic Use in a Neonatal Intensive Care Unit Practicing Integrative Medicine-A Retrospective Analysis. J Integr Complement Med. 2024 Apr;30(4):394-402. doi: 10.1089/jicm.2023.0001. Epub 2023 Oct 9. PMID 37815790